CLINICAL TRIAL: NCT00269971
Title: A Parallel Group Placebo-Controlled Study to Determine an Effective Dose Regimen for EPREX� (Epoetin Alfa) Sterile Solution to Reduce Transfusion Requirements in Patients Undergoing Major Elective Orthopedic Surgery
Brief Title: A Study to Determine an Effective Dose of Epoetin Alfa to Decrease the Number of Units of Blood Required to be Transfused During Hip Replacement Surgery.
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Ortho Inc., Canada (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005908
Record Dates: First submitted 2005-12-22; First posted 2005-12-26 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2011-09

CONDITIONS: Anemia; Blood Transfusion; Orthopedic Surgery
Keywords: hip replacement; hip replacement surgery; surgery; anemia; transfusions; blood; blood transfusions
MeSH Terms: conditions — Anemia | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: epoetin alfa

SUMMARY:
The purpose of this study is to determine an effective dose of epoetin alfa to be administered prior to surgery, to decrease the need for blood transfusions during hip replacement. Epoetin alfa is a genetically engineered protein that stimulates red blood cell production.

DETAILED DESCRIPTION:
Major surgical procedures may require blood transfusions both during and after the operation. Agents that can increase the rate of red blood cell production would reduce the need for blood transfusions. Epoetin alfa is a genetically engineered form of a natural hormone, erythropoietin, that stimulates red blood cell production. This is a randomized, double-blind, multicenter study in patients scheduled for first time hip replacement surgery. The study compares the effectiveness of 2 different doses of epoetin alfa (20,000 units or 40,000 units per week) for reducing the need for blood transfusions during the surgery. Eligible patients will be randomly assigned to one of three treatment groups: epoetin alfa 20,000 units per week, epoetin alfa 40,000 units per week, or placebo. Patients will be treated with study medication once a week for 4 weeks before their scheduled surgery. Effectiveness will be determined by the number of transfusions required during surgery. Other factors that determine effectiveness will be: the level of hemoglobin (the oxygen-carrying component of red blood cells) and the percentage of red blood cells in the patient's blood (hematocrit) prior to surgery; the number of developing red blood cells (reticulocytes); the iron stores in the patient's blood prior to surgery; the patient's quality of life after the surgery; and the time that elapses after surgery before the patient is discharged from the hospital. Safety evaluations will include the incidence of blood clots in the deep veins, the incidence and severity of other adverse events, and changes in clinical laboratory tests, vital signs, and physical examination findings throughout the study. The study hypothesis is that patients treated with epoetin alfa before hip replacement surgery will require fewer blood transfusions during the surgery compared with patients treated with placebo, and that the lower epoetin alfa dose (20,000 units per week) is as effective as the higher epoetin alfa dose (40,000 units per week). Patients will receive 20,000 units or 40,000 units of epoetin alfa injected under the skin once weekly for 4 weeks, or a matching placebo injection containing human serum albumin.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for first-time hip replacement surgery
* having no major medical conditions
* having a hemoglobin level of 98 - 137 grams per liter
* having adequate iron stores
* not participating in a self-donated blood program

Exclusion Criteria:

* Patients with a history of rheumatoid arthritis, blood disorders, recent bleeding episodes or an iron deficiency
* or having a history of seizures or uncontrolled high blood pressure (diastolic blood pressure > 100 mmHg)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 1996-05; Study Completion 1999-04 (Actual)

PRIMARY OUTCOMES:
Transfusion requirements at the time of surgery; hemoglobin and hematocrit levels, reticulocyte count, and iron stores prior to surgery; time to hospital discharge after surgery, and the patient's quality of life after surgery.

SECONDARY OUTCOMES:
Deep-vein blood clots; other adverse events, changes in clinical laboratory tests, vital sign measurements, and physical examination findings.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Ortho Inc. Clinical Trial, Study Director — Janssen-Ortho Inc., Canada

REFERENCES:
- See also: A study to determine an effective dose of epoetin alfa to decrease the number of units of blood required to be transfused for hip replacement surgery. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=364&filename=CR005908_CSR.pdf